CLINICAL TRIAL: NCT03816865
Title: Fibrosis, Inflammation and Brain Health in Atrial Fibrillation. The Norwegian Atrial Fibrillation and Stroke Study
Brief Title: Fibrosis, Inflammation and Brain Health in Atrial Fibrillation.
Acronym: NOR-FIB2
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Senior Consultant in Neurology, Oslo University Hospital
Other Study IDs: NOR-FIB2
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protocol synopsis Sponsor: Oslo University Hospital Title: Fibrosis, inflammation and cerebral infarction in patients with atrial fibrillation Study Design: The study is an observational prospective study of atrial fibrillation patients undergoing direct-current cardioversion.

Primary Objective: To assess the prevalence and causes of new silent cerebral ischemic lesions after programmed direct-current cardioversion using diffusion-weighted sequences in brain MRI (DWMRI).

Secondary Objectives:

To study the impact of inflammation measured by biomarkers and cardiac 18F-FDG-PET on the risk for new silent cerebral ischemic lesions after direct-current cardioversion for AF.

To assess the impact of fibrosis measured by biomarkers on the risk for new silent cerebral ischemic lesions after direct-current cardioversion for AF.

To assess cognitive and cerebral structural and metabolic changes after direct-current cardioversion for AF using cognitive assessments and cerebral and cardiac 18F-FDG-PET before and 12 months after treatment.

Number of Subjects: 50

Study Centers: Østfold Hospital Trust

Duration of Study Participation:

* Enrollment: 18 months
* Follow-up period: 12 months
* Total Study Duration: 30 months

Primary Endpoints:

• Number of new small cerebral infarcts detected with DWMRI two weeks after direct current cardioversion.

Secondary Endpoints:

* Rate of AF recurrence within 1 year after direct current cardioversion
* Change in levels of inflammation biomarkersfrom baseline to 12 months follow-up
* Change in levels of fibrosis biomarkers from baseline to 12 months follow-up
* Cognitive function at 12 months follow-up
* Changes in uptake pattern on cerebral 18F-FDG-PET from baseline to 12 months follow-up
* Changes in uptake pattern on cardiac 18F-FDG-PET from baseline to 12 months follow-up
* Brain volume at 12 months follow-up
* White matter volume 12 months follow-up
* Grey matter volume 12 months follow-up
* Cortical volume 12 months follow-up
* RSI-derived diffusion parameters 12 months follow-up: fast apparent diffusion coefficient, extracellular water fraction, fractional anisotropy; free water fraction; intracranial volume; NAWM: normal appearing white matter; neurite density; RSI: restriction spectrum imaging; sADC: slow apparent diffusion coefficient;restricted fractional anisotropy; white matter lesions.

ELIGIBILITY:
1. Known atrial fibrillation
2. Age <80 years
3. CHA2DS2-VASc ≤ 4
4. Planned direct-current cardioversion

Exclusion criteria:

1. CHA2DS2-VASc >4
2. Life expectancy less than 1 year
3. Patient otherwise not eligible for the study or adherent for follow-up (eg nonresident) or has concurrent disease affecting outcome (e.g. multiple sclerosis, cancer)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation undergoing direct-current cardioversion
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Number of new small cerebral infarcts detected with DWMRI two weeks after direct current cardioversion. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Østfold Hospital, Sarpsborg

IPD SHARING:
Plan to Share IPD: No